CLINICAL TRIAL: NCT03862911
Title: Phase III Randomized Controlled Trial and Economic Evaluation of Stereotactic Ablative Radiotherapy for Comprehensive Treatment of Oligometastatic (1-3 Metastases) Cancer (SABR-COMET-3)
Brief Title: Stereotactic Ablative Radiotherapy for Comprehensive Treatment of Oligometastatic (1-3 Metastases) Cancer
Acronym: SABR-COMET-3
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: British Columbia Cancer Agency (Other)
Collaborators: London Regional Cancer Program, Canada (Other); The Alfred (Other); Beacon Hospital, Ireland (Unknown); Cancer Trials Ireland (Network); Cancer Research UK Edinburgh Centre (Unknown); Bon Secours Cork Cancer Centre (Unknown); UPMC Hillman Cancer Centre (Unknown); Beatson West of Scotland Cancer Centre (Unknown); Tom Baker Cancer Centre (Other); Walker Family Cancer Centre (Unknown); Riverina Cancer Care Centre (Unknown); Aberdeen Royal Infirmary (Other)
Responsible Party: Principal Investigator, Robert Olson, Radiation Oncologist & Department Head Radiation Oncology & Developmental Radiotherapeutics, British Columbia Cancer Agency
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SABR-COMET-3
Record Dates: First submitted 2019-02-08; First posted 2019-03-05 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Metastatic Tumors
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Intervention Model Description: This study is a phase III multicentre randomized trial. Subjects will be randomized in a 1:2 ratio between current standard of care treatment (Arm 1) vs. standard of care treatment + SABR (Arm 2) to sites of known disease.
  Subjects will be stratified by two of the strongest prognostic factors, based on a large multi-institutional analysis: histology (Group 1: prostate, breast, or renal; Group 2: all others), and disease-free interval (defined as time from diagnosis of primary tumor until first detection of the metastases being treated on this trial; divided as ≤2 years vs >2 years).
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of Care Treatment (Arm 1) (Active Comparator): Standard of care, palliative radiotherapy, and chemotherapy at the discretion of the treating medical oncologist
  Interventions: Radiation: palliative radiotherapy
- Stereotactic Arm (Arm 2) (Experimental): Stereotactic ablative radiotherapy, and chemotherapy at the discretion of the treating medical oncologist
  Interventions: Radiation: Stereotactic ablative radiotherapy

INTERVENTIONS:
Radiation: palliative radiotherapy — Radiotherapy for patients in the standard arm should follow the principles of palliative radiotherapy as per the individual institution, with the goal of alleviating symptoms or preventing imminent complications. Patients in this arm should not receive stereotactic doses or radiotherapy boosts. Recommended dose fractionations in this arm will include 8 Gy in 1 fractions, 20 Gy in 5 fractions, and 30 Gy in 10 fractions.
  Arms: Standard of Care Treatment (Arm 1)
Radiation: Stereotactic ablative radiotherapy — Lung: Tumors 5 cm or less surrounded by lung parenchyma 48 Gy/4#, or 54 Gy/3#, daily or every second day Within 2 cm of mediastinum or brachial plexus 60 Gy/8#, daily
  Bone: Any bone 35 Gy/5#, or 24 Gy/2#, daily
  Brain: Stereotactic lesions (no whole brain RT) <2cm 20-24 Gy/1#, once 2-3 cm 18 Gy/1#, once Metastases only: 35Gy/5# to PTV, daily Whole brain + Mets: 35Gy to metastases, daily 20 Gy whole brain, daily
  Liver: 54 Gy/3#, every second day
  Adrenal/Pancreas: 40 Gy/5# / 35Gy/7#, daily
  Lymph Node: 40 Gy/5#, daily
  Arms: Stereotactic Arm (Arm 2)

SUMMARY:
Stereotactic Ablative Radiotherapy (SABR) is a modern RT technique that delivers high doses of radiation to small tumor targets using highly conformal techniques. SABR is non-invasive and delivered on an outpatient basis. The purpose of this study is to compare the effect of SABR, relative to standard of care (SOC) alone, on overall survival, progression-free survival, toxicity, and quality of life. An integrated economic evaluation will determine the cost per quality of life year gained using SABR (vs. SOC) and a translational component will enable identification of predictive/prognostic biomarkers of the oligometastatic state.

DETAILED DESCRIPTION:
TREATMENT PLAN

5.1.1 Standard Arm (Arm 1)

Radiotherapy for patients in the standard arm should follow the principles of palliative radiotherapy as per the individual institution, with the goal of alleviating symptoms or preventing imminent complications. Patients in this arm should not receive stereotactic doses or radiotherapy boosts. Recommended dose fractionations in this arm will include 8 Gy in 1 fractions, 20 Gy in 5 fractions, and 30 Gy in 10 fractions.

Systemic therapy will be pre-specified based on the standard of care approach for that patient, and it may include systemic therapy (cytotoxic, targeted, hormonal, or immunotherapy) or observation.

5.1.2 Experimental Arm (Arm 2)

Dose/Fractionation

Treatment recommendations are as follows:

Lung: Tumors 5 cm or less surrounded by lung parenchyma: 48 Gy in 4 fractions (12 Gy/#), 54 Gy in 3 fractions (18 Gy/#), daily or every second day

Lung: Within 2 cm of mediastinum or brachial plexus 60 Gy in 8 fractions (7.5 Gy/#) daily

Bone: Any bone 35 Gy in 5 fractions (7 Gy/#), 24 Gy in 2 fractions (12 Gy/#), daily

Brain: Stereotactic lesions (no whole brain RT):

<2cm 20-24 Gy in 1 fraction (20-24 Gy/#) Once

2-3 cm 18 Gy in 1 fraction (18 Gy/#) Once

3-4cm 15 Gy in 1 fraction (15 Gy/#) Once

Metastases only: 35Gy 5 7 Gy to PTV Daily, Whole brain + Mets: 35Gy to metastases 5 7 Gy to PTV Daily, 20 Gy whole brain 4 Gy WBRT Daily,

Liver: 54 Gy in 3 fractions (18 Gy/#), every second day

Adrenal/Pancreas: 40 Gy in 5 fractions (8 Gy/#)/ 35Gy in 5 fractions (7 Gy/#), daily

Lymph Node: 40 Gy in 5 fractions (8 Gy/#), daily

5.1.2.1 Immobilization Treatment will be setup using reproducible positioning and verified using an on-line protocol for all patients in this study. Immobilization may include a custom immobilization device, such as thermoplastic shell or vacuum bag, as per individual institutional practice when delivering SABR. Some centers do not use immobilization devices and have demonstrated high degrees of accuracy; this is acceptable in this study.

5.1.2.2 Imaging/Localization/Registration All patients in Arm 2 will undergo planning CT simulation. 4-dimensional CT will be used for tumors in the lungs, liver, or adrenals. Axial CT images will be obtained throughout the region of interest. For centres using stereotactic radiosurgery platforms, real-time tumor tracking and orthogonal imaging systems are permitted.

5.1.2.3 4D-CT Procedures

For patients undergoing 4D-CT, physics will review the 4D-CT images and will perform the following quality assurance procedures indicated on the 4D-CT template designed specifically for SABR:

i) Ensure all end inspiration (0%) tags exist and are in the right place. This ensures image integrity.

ii) If the quality of the 4D-CT images is not sufficient (determined by Physics), then standard 3D-CT will be performed on the fast helical CT or Untagged Average CT.

iii) Motion measurements in all 3 directions are performed:

1. If the motion is less than or equal to 7 mm and the good quality images exist, then treatment planning may be performed on the Untagged Average CT with the 50% or 60% phase (End Expiration) and the 0% phase being fused to it. This will define the IGTV.
2. If the motion is greater than 7 mm in any one direction, then respiratory-gated radiotherapy can be considered. In this case, treatment planning will be performed on a subset average CT dataset (usually labeled either 30%-60% Avg CT or 40%-70% Avg CT) generated by Physics. This is an average CT over the intended gated interval. Therefore, the GTV that is delineated on this scan will incorporate residual motion in the intended gated interval. The 0% phase will also be fused to this dataset. The PTV for planning will include the GTV delineated on the subset average CT plus margins for microscopic extension (Physician's discretion) and setup uncertainty. The GTV_0% should also be delineated and combined with the GTV delineated on the subset average CT to define an additional volume labeled IGTV_CBCT. This contour may be used for image registration with CBCT only.

5.1.2.4 Volume Definitions (Arm 2) For all lesions, the gross tumor volume (GTV) will be defined as the visible tumor on CT and/or MRI imaging +/- PET. No additional margin will be added for microscopic spread of disease (i.e. Clinical Target Volume [CTV]=GTV). For bone lesions, CTV of 3-5mm will be allowed. For vertebral lesions, anatomic approach will be taken as per International Spinal consortium guideline (Cox 2012)

An anatomic approach is taken to the CTV based on where the disease within the spinal segment is located. The rules for CTV are as follows:

1. If the vertebral body is involved with GTV then the entire vertebral body is taken as CTV.
2. If the ipsilateral pedicle and/or transverse process has GTV then the entire ipsilateral posterior segment (pedicle, lamina and transverse process) ±the spinous process is taken into the CTV. The inclusion of the spinous process is per the discretion of the radiation oncologist.
3. If the ipsilateral pedicle, lamina, and/or transverse process has GTV, then the entire ipsilateral posterior segment (pedicle, lamina, and transverse process) plus the spinous process is taken into the CTV
4. If bilateral involvement of the pedicle and/or transverse process with GTV, then the posterior segment anatomy ± the spinous process is taken into the CTV. The inclusion of the spinous process is per the discretion of the radiation oncologist.
5. If bilateral involvement of the pedicles and lamina, and/or transverse process with GTV, then the entire posterior segment anatomy is taken into the CTV, including the spinous process.
6. If the spinous process is involved with GTV alone then the bilateral lamina ± pedicles are to be taken into the CTV.

The International Spinal Consortium Guideline is a reference for CTV delineation (Cox 2012) and can be adhered to as described.

In the case of epidural disease, a 5 mm anatomic margin (excluding the spinal cord) beyond the GTV may be used within the epidural compartment including in the cranio-caudal direction. A circumferential CTV as per a donut based CTV is allowed and encouraged in the case of epidural disease at the discretion of the treating radiation oncologist. If paraspinal disease present, a minimum 5 mm CTV margin may be applied beyond the GTV.

A Planning Target Volume (PTV) margin of 2-5 mm will be added depending on site of disease, immobilization, and institutional set-up accuracy: 2-3 mm margins should be used for spinal stereotactic treatments, 0-2 mm for brain tumors, and 5 mm for other sites.

Targets should be named based on the organ involved, and numbered from cranially to caudally. For example, in a patient with 3 lung lesions, there would be: GTV_lung_1, GTV_lung_2, and GTV_lung_3, and corresponding PTV_lung_1, PTV_lung_2_, and PTV_lung_3, representing the lesions from superior to inferior.

For spinal lesions, a pre-treatment MRI is required to assess the extent of disease and position of the cord. This must be fused with the planning CT scan. A Planning Organ at Risk Volume (PRV) expansion of 2 mm will be added to the spinal cord, and dose constraints for the spinal cord apply to this PRV. Alternatively, the thecal sac may be used as the PRV. For radiosurgery platforms, a PRV margin of 1 mm is permitted for the spinal cord.

Organ At Risk (OAR) Doses OAR doses are listed in Appendix 1 of protocol. OAR doses may not be exceeded except in the case of chestwall / ribs. In cases where the PTV coverage cannot be achieved without exceeding OAR doses, the PTV coverage is to be compromised. All serial organised OARs within 5 cm of the PTV must be contoured (partial organ contours allowed); for parallel organised organs (liver, lung, etc.) within 5cm of PTV, the whole organs need to be contoured. This should be tested for each PTV by creating a 5 cm expansion to examine which OARs lie within that expansion.

Treatment Planning Treatment can be delivered using static beams (either 3D-conformal radiotherapy or intensity-modulated) or rotational therapy (volumetric modulated arc therapy, or tomotherapy).

Dose constraints may not be exceeded (except chestwall/ribs). If a dose constraint cannot be achieved due to overlap of the target with an organ at risk, the fractionation can be increased or the target coverage compromised in order to meet the constraint. In cases where the target coverage or dose must be reduced, the priority for dose coverage is the GTV (e.g. attempt to cover as much of the GTV as possible with the prescription dose). All such cases of dose reduction or target coverage compromise must be approved by the local PI prior to treatment. For vertebral tumors, note that the spinal cord constraints apply to the PRV (see section 6.2.5).

For all targets, doses should be prescribed to 60-90% isodose line surrounding the PTV, and all hotspots should fall within the GTV. 95% of the PTV should be covered by the prescription dose, and 99% of the PTV should be covered by 90% of the prescription dose.

Doses must be corrected for tissue inhomogeneities. Several non-overlapping 6/10 MV beams (on the order of 7-11 beams) or 1-2 VMAT arcs combined possibly with a few non-coplanar beams should be utilized. Non-coplanar beams can be used to reduce 50% isodose volume.

The number of isocentres is at the discretion of the treating physician, physicists, and dosimetrists. Generally, metastases can be treated with separate isocenters if they are well-separated.

The scheduling and sequence of treating each metastasis is at the discretion of individual physicians, but in general should begin with the brain, due to risks associated with progression. All SABR must be completed within 2 weeks.

5.1.2.5 Quality Assurance (Arm 2)

In order to ensure patient safety and effective treatment delivery, a robust quality assurance protocol is incorporated. The following requirements must be completed for each patient:

* Prior to treatment, each patient must be discussed at quality assurance (QA) rounds or be peer reviewed by a radiation oncologist with SABR expertise.
* All radiotherapy plans must meet target dose levels for organs at risk (except chestwall/ribs) (Appendix 1). Prior to plan approval, the dose to each organ at risk must be verified by the physicist or treating physician.
* All dose delivery for intensity-modulated plans (including arc-based treatments) will be confirmed before treatment by physics staff.

5.1.2.6 Systemic Therapy Patients treated with prior systemic therapy are eligible for this study, however, no chemotherapy agents (cytotoxic, or molecularly targeted agents) are allowed within the period of time commencing 2 weeks prior to radiation lasting until 1 week after the last fraction. Hormonal therapy is allowed. Use of chemotherapy schemes containing potent enhancers of radiation damage (e.g. gemcitabine, adriamycin/doxorubicin, bevacizumab) are discouraged within the first month after radiation.

5.1.2.7 Further radiotherapy for progressive disease at new metastatic sites Patients in Arm 1 who develop new, untreated metastatic deposits should be treated with standard-of-care approaches. SABR to those sites is not permitted, except for unique scenarios where it would be considered standard of care (e.g. all disease controlled on systemic therapy with a newly developed brain metastasis). Apart from brain metastases, treatment of 'oligo-progression' with SABR is not permitted.

Patients in Arm 2 who develop new, untreated metastatic deposits should be considered for SABR at those sites, if such deposits can be treated safely with SABR, and if the treating institution offers SABR for that body site. If SABR is not possible, then palliative RT can be delivered if indicated.

5.1.2.8 Quality Assurance for Centres Joining Study Prior to opening the study, each participating research centre will be required to send to one of the Principal Investigators a mock treatment plan for the anatomic sites that will be treated (e.g. Lung, brain, liver, adrenal), to ensure that the treatment plans are designed in compliance with the protocol. The principal investigators will provide pertinent CT datasets. Each participating research centre can choose which tumor sites will be treated at their individual centre (i.e. some centres may only choose to treat a subset of the eligible metastatic sites). Sites that have prior accreditation for SABR through a clinical trial (e.g. SABR-COMET, or organ-specific SABR trials) are exempt from this requirement for the organ sites that have been accredited in those trials.

ELIGIBILITY:
Inclusion Criteria:

* Total number of 1-3 current metastases, and a maximum 8 lifetime metastases
* Age 18 or older
* Willing to provide informed consent
* ECOG score 0-2
* Life expectancy >6 months
* Histologically confirmed malignancy with metastatic disease detected on imaging. Biopsy of metastasis is preferred, but not required.
* Controlled primary tumor

  * defined as: at least 3 months since original tumor treated definitively, with no progression at primary site (can be considered controlled if no evidence of the primary tumour on imaging)
* A history and physical exam, including ECOG performance status, performed within 6 weeks prior to trial enrollment
* Not suitable for resection at all sites or decline surgery
* Patient has had a CT chest, abdomen and pelvis or PET-CT within 8 weeks prior to enrollment, and within 12 weeks prior to treatment(if randomized to SABR). CT neck as clinically indicated.
* Patient has had a nuclear bone scan (if no PET-CT) within 8 weeks prior to enrollment, and within 12 weeks prior to treatment(if randomized to SABR)
* If solitary lung nodule for which biopsy is unsuccessful or not possible, patient has had an FDG PET scan or CT (chest, abdomen, pelvis) and bone scan within 8 weeks prior to enrollment, and with 12 weeks prior to treatment (if randomized to SABR). CT neck as clinically indicated.
* If colorectal primary with rising CEA, but equivocal imaging, patient has had an FDG PET scan within 8 weeks prior to enrollment, and within 12 weeks prior to treatment(if randomized to SABR)
* Patient has had CT or MRI brain imaging if primary has a propensity for CNS metastasis within 8 weeks prior to enrollment, and within 12 weeks prior to treatment(if randomized to SABR)
* Patient is judged able to:
* Maintain a stable position during therapy
* Tolerate immobilization device(s) that may be required to deliver SABR safely
* Negative pregnancy test for Women of Child-Bearing potential (WOCBP) within 4 weeks of RT start date
* Patient is able and willing to complete the quality of life questionnaires, and other assessments that are a part of this study, via paper or online using REDCap (if email address is provided by participant on the informed consent)

Waivers to the inclusion criteria will NOT be allowed.

Exclusion Criteria:

* Lesion in femoral bone requiring surgical fixation
* Chemotherapy agents (cytotoxic, or molecularly targeted agents) used within the period of time commencing 2 weeks prior to radiation, lasting until 1 week after the last fraction for patients randomized to SABR
* Serious medical comorbidities precluding radiotherapy. These include interstitial lung disease in patients requiring thoracic radiation, Crohn's disease in patients where the GI tract will receive radiotherapy, and connective tissue disorders such as lupus or scleroderma.
* Substantial overlap with a previously treated radiation volume. Prior radiotherapy in general is allowed, as long as the composite plan meets dose constraints herein. For patients treated with conventional radiation previously, biological effective dose calculations should be used to equate previous doses to the tolerance doses listed below. All such cases should be discussed with one of the study PIs.
* Concurrent malignant cancer, or history of malignant cancers within the past 5 years
* Malignant pleural effusion
* History of poor lung function (if treating near lung)
* History of poor liver function (if treating near liver)
* Inability to treat all sites of disease
* Maximum size of 5 cm for lesions outside the brain, except:

  * Bone metastases over 5 cm may be included, if in the opinion of the local PI it can be treated safely (e.g. rib, scapula, pelvis)
  * Any brain metastasis >3 cm in size or a total volume of brain metastases greater than 30 cc.
* Clinical or radiologic evidence of spinal cord compression, or epidural tumor within <2 mm of the spinal cord. Patients can be eligible if surgical resection has been performed, but the surgical site counts toward the total of up to 8 lifetime metastases.
* Dominant brain metastasis requiring surgical decompression
* Pregnant or breastfeeding women

Waivers to exclusion criteria will NOT be allowed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2019-11-01 (Actual); Primary Completion 2030-11-24 (Estimated); Study Completion 2030-12-31 (Estimated)

PRIMARY OUTCOMES:
Overall survival | At approximately end of year 5 (study completion)
  Time from randomization to death from any cause

SECONDARY OUTCOMES:
Side effects | At 6 weeks, 3 months, 6 months, and every 6 months post treatment for years 1 and 2. At approximately end of years 3, 4, and 5.
  Occurrences of grade 2 or higher adverse events
Progression-free survival (PFS) | At 6 weeks, 3 months, 6 months, and every 6 months post treatment for years 1 and 2. At approximately end of years 3, 4, and 5.
  Time from randomization to disease progression at any site or death.
Patient-reported quality of life (QoL) | At baseline, 6 weeks, 3 months, 6 months, and every 6 months post treatment for years 1 and 2. At approximately end of years 3, 4, and 5.
  Functional Assessment of Cancer Therapy- General (FACT-G) questionnaire
Health-related quality of life (HRQoL) questionnaire | At baseline, 3 months, 6 months, and every 6 months post treatment for years 1 and 2. At approximately end of years 3, 4, and 5.
  EuroQOL Group EQ-5D-5L
Resource Utilization (Patient and Provider Reported) | At 3 months, 6 months, and every 6 months post treatment for years 1 and 2. At approximately end of years 3, 4, and 5.
  Number of hospital admissions, ER visits, systemic or radiation therapy
Correlation between candidate biomarkers of oligometastatic disease (blood-derived) and oncologic outcomes | At baseline, 3 months, and disease progression or study completion (Year 5)
  CTC and ctDNA Enumeration

CONTACTS AND LOCATIONS:
Overall Officials: Robert A Olson, MD, MSc, FRCPC, Principal Investigator — BC Cancer Prince George
Locations (17):
- Australia (3):
  - Cancer Care Griffith, Griffith, New South Wales
  - Riverina Cancer Care Centre, Wagga Wagga, New South Wales
  - Alfred Hospital, Melbourne, Victoria
- Canada (8):
  - Tom Baker Cancer Centre/Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - BC Cancer, Kelowna, British Columbia
  - BC Cancer - Prince George, Prince George, British Columbia
  - BC Cancer, Surrey, British Columbia
  - BC Cancer, Vancouver, British Columbia
  - BC Cancer, Victoria, British Columbia
  - London Health Sciences Centre, London, Ontario
  - Walker Family Cancer Centre, Saint Catharines, Ontario
- Ireland (3):
  - St. Luke's Radiation Oncology Network, Rathgar, Dublin
  - Beacon Hospital, Dublin, Sandyford
  - Bon Secours Radiotherapy Cork in partnership with UPMC Hillman Cancer Centre, Cork
- United Kingdom (3):
  - Aberdeen Royal Infirmary, Aberdeen, Scotland
  - Edinburgh Cancer Centre, Edinburgh, Scotland
  - Beatson West of Scotland Cancer Centre, Glasgow

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Hellman S, Weichselbaum RR. Oligometastases. J Clin Oncol. 1995 Jan;13(1):8-10. doi: 10.1200/JCO.1995.13.1.8. No abstract available. PMID 7799047
- [Background] Pastorino U, Buyse M, Friedel G, Ginsberg RJ, Girard P, Goldstraw P, Johnston M, McCormack P, Pass H, Putnam JB Jr; International Registry of Lung Metastases. Long-term results of lung metastasectomy: prognostic analyses based on 5206 cases. J Thorac Cardiovasc Surg. 1997 Jan;113(1):37-49. doi: 10.1016/s0022-5223(97)70397-0. PMID 9011700
- [Background] Hong JC, Ayala-Peacock DN, Lee J, Blackstock AW, Okunieff P, Sung MW, Weichselbaum RR, Kao J, Urbanic JJ, Milano MT, Chmura SJ, Salama JK. Classification for long-term survival in oligometastatic patients treated with ablative radiotherapy: A multi-institutional pooled analysis. PLoS One. 2018 Apr 12;13(4):e0195149. doi: 10.1371/journal.pone.0195149. eCollection 2018. PMID 29649281
- [Background] Primrose J, Treasure T, Fiorentino F. Lung metastasectomy in colorectal cancer: is this surgery effective in prolonging life? Respirology. 2010 Jul;15(5):742-6. doi: 10.1111/j.1440-1843.2010.01759.x. Epub 2010 Apr 23. PMID 20456671
- [Background] Palma DA, Salama JK, Lo SS, Senan S, Treasure T, Govindan R, Weichselbaum R. The oligometastatic state - separating truth from wishful thinking. Nat Rev Clin Oncol. 2014 Sep;11(9):549-57. doi: 10.1038/nrclinonc.2014.96. Epub 2014 Jun 24. PMID 24958182
- [Background] Iyengar P, Wardak Z, Gerber DE, Tumati V, Ahn C, Hughes RS, Dowell JE, Cheedella N, Nedzi L, Westover KD, Pulipparacharuvil S, Choy H, Timmerman RD. Consolidative Radiotherapy for Limited Metastatic Non-Small-Cell Lung Cancer: A Phase 2 Randomized Clinical Trial. JAMA Oncol. 2018 Jan 11;4(1):e173501. doi: 10.1001/jamaoncol.2017.3501. Epub 2018 Jan 11. PMID 28973074
- [Background] Gomez DR, Blumenschein GR Jr, Lee JJ, Hernandez M, Ye R, Camidge DR, Doebele RC, Skoulidis F, Gaspar LE, Gibbons DL, Karam JA, Kavanagh BD, Tang C, Komaki R, Louie AV, Palma DA, Tsao AS, Sepesi B, William WN, Zhang J, Shi Q, Wang XS, Swisher SG, Heymach JV. Local consolidative therapy versus maintenance therapy or observation for patients with oligometastatic non-small-cell lung cancer without progression after first-line systemic therapy: a multicentre, randomised, controlled, phase 2 study. Lancet Oncol. 2016 Dec;17(12):1672-1682. doi: 10.1016/S1470-2045(16)30532-0. Epub 2016 Oct 24. PMID 27789196
- [Background] Ruers T, Van Coevorden F, Punt CJ, Pierie JE, Borel-Rinkes I, Ledermann JA, Poston G, Bechstein W, Lentz MA, Mauer M, Folprecht G, Van Cutsem E, Ducreux M, Nordlinger B; European Organisation for Research and Treatment of Cancer (EORTC); Gastro-Intestinal Tract Cancer Group; Arbeitsgruppe Lebermetastasen und tumoren in der Chirurgischen Arbeitsgemeinschaft Onkologie (ALM-CAO); National Cancer Research Institute Colorectal Clinical Study Group (NCRI CCSG). Local Treatment of Unresectable Colorectal Liver Metastases: Results of a Randomized Phase II Trial. J Natl Cancer Inst. 2017 Sep 1;109(9):djx015. doi: 10.1093/jnci/djx015. PMID 28376151
- [Background] Ruers T, Punt C, Van Coevorden F, Pierie JPEN, Borel-Rinkes I, Ledermann JA, Poston G, Bechstein W, Lentz MA, Mauer M, Van Cutsem E, Lutz MP, Nordlinger B; EORTC Gastro-Intestinal Tract Cancer Group; Arbeitsgruppe Lebermetastasen und-tumoren in der Chirurgischen Arbeitsgemeinschaft Onkologie (ALM-CAO) and the National Cancer Research Institute Colorectal Clinical Study Group (NCRI CCSG). Radiofrequency ablation combined with systemic treatment versus systemic treatment alone in patients with non-resectable colorectal liver metastases: a randomized EORTC Intergroup phase II study (EORTC 40004). Ann Oncol. 2012 Oct;23(10):2619-2626. doi: 10.1093/annonc/mds053. Epub 2012 Mar 19. PMID 22431703
- [Background] Cheruvu P, Metcalfe SK, Metcalfe J, Chen Y, Okunieff P, Milano MT. Comparison of outcomes in patients with stage III versus limited stage IV non-small cell lung cancer. Radiat Oncol. 2011 Jun 30;6:80. doi: 10.1186/1748-717X-6-80. PMID 21718501
- [Background] Rava P, Leonard K, Sioshansi S, Curran B, Wazer DE, Cosgrove GR, Noren G, Hepel JT. Survival among patients with 10 or more brain metastases treated with stereotactic radiosurgery. J Neurosurg. 2013 Aug;119(2):457-62. doi: 10.3171/2013.4.JNS121751. Epub 2013 May 10. PMID 23662828
- [Background] Ritter TA, Matuszak M, Chetty IJ, Mayo CS, Wu J, Iyengar P, Weldon M, Robinson C, Xiao Y, Timmerman RD. Application of Critical Volume-Dose Constraints for Stereotactic Body Radiation Therapy in NRG Radiation Therapy Trials. Int J Radiat Oncol Biol Phys. 2017 May 1;98(1):34-36. doi: 10.1016/j.ijrobp.2017.01.204. No abstract available. PMID 28587050
- [Background] De Oliveira C, Pataky R, Bremner KE, Rangrej J, Chan KK, Cheung WY, Hoch JS, Peacock S, Krahn MD. Estimating the Cost of Cancer Care in British Columbia and Ontario: A Canadian Inter-Provincial Comparison. Healthc Policy. 2017 Feb;12(3):95-108. PMID 28277207
- [Background] Devlin NJ, Krabbe PF. The development of new research methods for the valuation of EQ-5D-5L. Eur J Health Econ. 2013 Jul;14 Suppl 1(Suppl 1):S1-3. doi: 10.1007/s10198-013-0502-3. No abstract available. PMID 23900659
- [Background] Leggett LE, Khadaroo RG, Holroyd-Leduc J, Lorenzetti DL, Hanson H, Wagg A, Padwal R, Clement F. Measuring Resource Utilization: A Systematic Review of Validated Self-Reported Questionnaires. Medicine (Baltimore). 2016 Mar;95(10):e2759. doi: 10.1097/MD.0000000000002759. PMID 26962773
- [Derived] Olson R, Mathews L, Liu M, Schellenberg D, Mou B, Berrang T, Harrow S, Correa RJM, Bhat V, Pai H, Mohamed I, Miller S, Schneiders F, Laba J, Wilke D, Senthi S, Louie AV, Swaminath A, Chalmers A, Gaede S, Warner A, de Gruijl TD, Allan A, Palma DA. Stereotactic ablative radiotherapy for the comprehensive treatment of 1-3 Oligometastatic tumors (SABR-COMET-3): study protocol for a randomized phase III trial. BMC Cancer. 2020 May 5;20(1):380. doi: 10.1186/s12885-020-06876-4. PMID 32370765

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-05-15): https://cdn.clinicaltrials.gov/large-docs/11/NCT03862911/Prot_SAP_010.pdf